CLINICAL TRIAL: NCT05793333
Title: Histological and Molecular Characteristics Predict the Risk of Nodal Involvement in Endometrial Cancer: a Prospective Study
Brief Title: Predictors of Node Positivity in Endometrial Cancer
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Valentina Chiappa, Dr, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: 142020
Record Dates: First submitted 2023-03-04; First posted 2023-03-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Cancer
Keywords: sentinel node; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To investigate the role of histological and moleculr profile of endometrial cancer patietns in predicting the risk of nodal metastases in endometrila cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed endometrila cancer
* Data on molecular genomic profiling (POLE mutated, p53 abnormalities, MMRd/MSI-H, and NSMP)
* Data on histological characteristics of the ttumor
* Execution of sentinel node mapping
* Data on sentinel node status (negative vs. positive)

Exclusion Criteria:

* Stage IVB endoemtrial cancer
* consent withdraw

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patietns were submitted to standard treatment modality for managing endometrial cancer. They will receive hsyterectomy (with or without bilateral salpingo-oophorectomy) plus sentinel ndoe mapping.
  After the procedures data regarding hystologcial charactersitcs of the tumor and molecular features will be analyzed (as routine cliical practice).
  We will correlate those data with findings achieved by sentinel nodes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
positive nodes | 12 months
  positive nodes detected by sentinel node mappinig

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Bogani, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogani G, Lalli L, Casarin J, Ghezzi F, Chiappa V, Fanfani F, Scambia G, Raspagliesi F. Predicting the Risk of nOdal disease with histological and Molecular features in Endometrial cancer: the prospective PROME trial. Int J Gynecol Cancer. 2024 Sep 2;34(9):1366-1372. doi: 10.1136/ijgc-2024-005416. PMID 38658017